CLINICAL TRIAL: NCT06375031
Title: Comparing Pharmacokinetics and Pharmacodynamics Between HR011408 and NovoRapid® in Subjects With Diabetics- A Randomized, Double-Blind, Three-cycle Crossover Phase I Clinical Trial
Brief Title: Comparison of HR011408 and NovoRapid® in Subjects With Diabetics
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: HR011408-103
Record Dates: First submitted 2024-04-16; First posted 2024-04-19 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus | interventions — Insulin Aspart

STUDY DESIGN:
Intervention Model Description: The study was designed as a multi-center, randomized, double-blind, three-cycle crossover, positive drug control (NovoRapid ®) To compare the pharmacokinetics, pharmacodynamics, safety, and tolerability of a single injection of HR011408 or NovoRapid ® before or after a standard meal test in patients with type 1 or type 2 diabetes.
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm 1: Medication regimen A-B-C (Experimental)
  Interventions: Drug: HR011408 injection; HR011408 injection Placebo; Drug: NovoRapid®; HR011408 injection Placebo; Drug: HR011408 injection Placebo; HR011408 injection
- Arm 2: Medication regimen B-C-A (Experimental)
  Interventions: Drug: HR011408 injection; HR011408 injection Placebo; Drug: NovoRapid®; HR011408 injection Placebo; Drug: HR011408 injection Placebo; HR011408 injection
- Arm 3: Medication regimen C-A-B (Experimental)
  Interventions: Drug: HR011408 injection; HR011408 injection Placebo; Drug: NovoRapid®; HR011408 injection Placebo; Drug: HR011408 injection Placebo; HR011408 injection

INTERVENTIONS:
Drug: HR011408 injection; HR011408 injection Placebo — Medication regimen-A:
  HR011408 injection, ante cibum; HR011408 injection Placebo , post cibum
Drug: NovoRapid®; HR011408 injection Placebo — Medication regimen-B:
  NovoRapid®, ante cibum; HR011408 injection Placebo, post cibum
Drug: HR011408 injection Placebo; HR011408 injection — Medication regimen-C:
  HR011408 injection Placebo, ante cibum:
  HR011408 injection, post cibum

SUMMARY:
The objective of the study is to compare the pharmacokinetics and pharmacodynamics between HR011408 and NovoRapid® in Subjects with Diabetics.

ELIGIBILITY:
Inclusion Criteria:

- Subjects had to meet all the following criteria to enrol this study

1. Male or female aged 18-64 years (both inclusive)；
2. Body mass index 18.5-35.0 kg/m2 (both inclusive)；
3. Diagnosed with type 1 diabetes or type 2 diabetes≥ 12 months at screening；
4. HbA1c ≤9.0% by local laboratory at screening；
5. Current treatment with any basal-bolus insulin regimen or continuous subcutaneous insulin infusion(CSII) for ≥ 8 weeks. Patients with type 2 diabetes can also take metformin but require a stable metformin dose for ≥8 weeks；
6. Current total daily insulin treatment < 1.2 U/kg/day, and total daily bolus insulin treatment ≥ 0.3 U/kg/day and < 0.7 U/kg/day.

Exclusion Criteria:

- Subjects who meet any of the following criteria will be excluded from this study.

1. The following laboratory or ancillary abnormalities were present from screening until randomization:

1) Poor blood pressure control, defined as systolic blood pressure ≥160 mmHg or diastolic blood pressure ≥100 mmHg.

2. Subject has any history or evidence meet the following diseases or conditions:

1. have had severe hypoglycaemia episodes within 6 months before screening as judged by the investigator.
2. Have hospitalization due to diabetic ketoacidosis or hyperglycaemic hyperosmolar state within 6 months prior to screening;
3. Proliferative retinopathy, maculopathy, and/or severe neuropathy, in particular autonomic neuropathy, as judged by the investigator.

3. Previous and anticipated concomitant treatments:

1. Not able or willing to refrain from any use of herbal products and non-routine vitamins within 14 days or within 5 half-lives (whichever is longer), and routine vitamins within 48 hours prior to trial product administration
2. Within 1 month or have within 5 half-lives (whichever is longer) participated in any trail (defined participate in trail as having had randomized) of using investigational drug or therapy prior to screening.

4. General information:

1. Smoker (defined as a subject who is smoking more than 5 cigarettes or the equivalent nicotine per day).
2. Previous participation in this study. Participation was defined as randomised.

5. Any other situation judged by investigator that may endanger the safety of the subjects or influence the evaluation of the results.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-05 (Estimated); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-07-15 (Estimated)

PRIMARY OUTCOMES:
Area under the serum concentration-time curve of insulin aspart | From 0 to 30 mins after trial product administration

SECONDARY OUTCOMES:
Area under the serum concentration-time curve of insulin aspart | From 0 to 6 hours after trial product administration
Plasma glucose concentration | From 0 to 6 hours after start of a standardised meal
Number of subjects with adverse events and severity of adverse events | From first dose to the last visit, approximately 2 months

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Hospital of Anhui Medical University, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: Undecided